CLINICAL TRIAL: NCT06746064
Title: A Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability and Pharmacokinetics of CHF10073 After Single and Multiple Ascending Doses in Healthy Volunteers Via Inhalation and the Effect of Multiple Doses of Itraconazole on CHF10073 Exposure
Brief Title: A Study to Investigate the Safety, Tolerability and Pharmacokinetics of Inhaled CHF10073 After Single and Multiple Doses in Healthy Volunteers and the Effect of Itraconazole on CHF10073 Exposure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CLI-010073AA1-01; 2024-515442-17-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-26; First posted 2024-12-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — Itraconazole

STUDY DESIGN:
Intervention Model Description: Part 1 - SAD (single ascending dose): Randomised, double-blind, placebo-controlled, single-dose escalation, parallel-group design in HVs.
  Part 2 - MAD (multiple ascending dose): Randomised, double-blind, placebo-controlled, repeated-dose escalation, parallel-group design in HVs; Part 3: Non-randomised, open-label, single dose design in HVs Part 4 - Non-randomised, open-label, one-sequence, two-period crossover design in HVs.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHF10073 active (Experimental)
  Interventions: Drug: CHF10073 (Part 1 - SAD); Drug: CHF10073 (Part 2 - MAD); Drug: CHF10073 (Part 3); Drug: CHF10073 (Part 4)
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo (Part 1 - SAD); Drug: Placebo (Part 2 - MAD)
- CHF10073 + itraconazole (Experimental)
  Interventions: Drug: itraconazole (Part 4); Drug: CHF10073 (Part 4)

INTERVENTIONS:
Drug: CHF10073 (Part 1 - SAD) — Single doses of CHF10073 for each cohort
  Arms: CHF10073 active
Drug: Placebo (Part 1 - SAD) — Single doses of placebo matching CHF10073 for each cohort
  Arms: placebo
Drug: CHF10073 (Part 2 - MAD) — Multiple doses of CHF10073 for each cohort
  Arms: CHF10073 active
Drug: CHF10073 (Part 3) — Single dose of CHF10073
  Arms: CHF10073 active
Drug: Placebo (Part 2 - MAD) — Multiple doses of placebo matching CHF10073 for each cohort
  Arms: placebo
Drug: itraconazole (Part 4) — Multiple dose of itraconazole in treatment period 2
  Arms: CHF10073 + itraconazole
Drug: CHF10073 (Part 4) — Single dose of CHF10073 in Treatment Period 1 and 2
  Arms: CHF10073 + itraconazole; CHF10073 active

SUMMARY:
The objective of this study is to assess the safety and tolerability of single ascending doses of inhaled CHF10073 (Part 1 of the study) and multiple ascending doses of CHF10073 (Part 2 of the study). The study will also evaluate the PK profile of study drug in plasma and urine after single and repeated administrations of CHF10073.

In addition, this study will also investigate the metabolites profile of CHF10073 in plasma, urine and faeces (Part 2 of the study) and the PK profile of CHF10073 in the lungs after bronchoalveolar lavage (BAL) (Part 3 of the study).

In addition, the effect of multiple doses of itraconazole on the pharmacokinetic profile of CHF10073 will be investigated (Part 4 of the study).

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent;
* Healthy male (Part 1 to 4) or female (Part 4) 18-55 years;
* Understanding of the study procedures and the correct use of the inhalers;
* BMI between 18.5 and 30.0 kg/m2;
* Non- or ex-smokers (<5 pack-years and stopped smoking >1 year prior to screening);
* Good physical and mental status;
* Vital signs within normal limits; body temperature <37.5°C;
* 12-lead digitised ECG in triplicate considered as normal;
* Lung function measurements within normal limits;
* Males with pregnant or non-pregnant women of childbearing potential (WOCBP) partners must be willing to use contraception
* Part 4 only: women of non-childbearing potential (WONCBP) or WOCBP with fertile male parters willing to use contraception

Exclusion Criteria:

* Recent participation in another clinical trial;
* Clinically significant abnormal 24h Holter ECG (Part 1 and 2);
* Clinically relevant and uncontrolled medical disorders ;
* Subjects with history of respiratory diseases ;
* Presence of any current or recent infection;
* Clinically relevant abnormal laboratory values;
* Abnormal liver enzymes;
* Positive results from the Hepatitis serology results;
* Positive HIV-1 or HIV-2 serology results ;
* Recent blood donation or blood loss (≥450 mL) ;
* Heavy caffeine drinker ;
* Recent use of any kind of electronic smoking devices;
* Documented history of alcohol abuse within 12 months prior to screening ;
* Documented history of drug abuse within 12 months prior to screening ;
* Intake of non-permitted concomitant medications ;
* Known intolerance and/or hypersensitivity to any of the study excipients ;
* Unsuitable veins for repeated venipuncture;
* Part 3 only: contraindication to the BAL procedure;
* Part 3 only: recent lower respiratory tract infections
* Part 4 only: known allergy to antifungal medicines;
* Part 4 and females only: pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 155 (Actual)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-02-04 (Actual); Study Completion 2026-02-04 (Actual)

PRIMARY OUTCOMES:
Adverse events and adverse drug reactions | Through study completion, around 8 weeks in Part 1, from 10 to 13 weeks in Part 2, for about 7-8 weeks in Part 3 and for about 15 up to 17 weeks in Part 4
Vital signs (Systolic and diastolic Blood Pressure) | From screening up to 42 days post-dose
Absolute Values for 12-lead Electrocardiogram (ECG) Recording of HR (heart rate), HR from 0 to 24 hours, hourly HR | From screening up to 28 days post-dose
Absolute Values for 12-lead ECGs Recording of Intervals | From screening up to 28 days post-dose
  Intervals recorded: PR, QRS, QT, QTcF
Change from Baseline for Post-dose 12-lead ECGs Recording of HR, HR from 0 to 24 hours, hourly HR | From screening up to 28 days post-dose
Change from Baseline for Post-dose 12-lead ECGs Recording of Intervals | From screening up to 28 days post-dose
  Intervals recorded: PR, QRS, QT, QTcF
Number and percentage of subjects with abnormal actual QTcF (Fridericia-corrected QT Interval). | Part 1 and 2 only: From screening up to 28 days post-dose
Number and percentage of subjects with abnormal change from the baseline of QTcF and HR from 0 to 24 hours | Part 1 and 2 only: From screening up to 28 days post-dose
Number of subjects and percentages by treatment with abnormal parameters derived from 24h Holter ECG recording (total pauses >2.5 secs, atrial fibrillation and atrial flutter, ventricular runs, PAC burden, PVC burden and aberrant morphologies) | Part 1 and 2 only: From screening up to 28 days post-dose
Number of subjects with abnormal blood laboratory test results | From screening up to 28 days post-dose
  Quantitative laboratory parameters (chemistry and haematology) will be summarised by treatment as absolute value and change from baseline using descriptive statistics.
Number of subjects with abnormal urine laboratory test results | From screening up to 28 days post-dose
Spirometry (FEV1 (Forced exhalation volume in the first second)) | From screening up to 28 days post-dose
Cough recording: percentage of days with cough episodes during the treatment period | Part 2 only: From first dosing up to 28 days post-dose
Cough recording: average VAS (visual analogue scale)) | Part 2 only: From first dosing up to 28 days post-dose
CHF10073 plasma AUCt (Area Under the Curve from time 0 to time t) | From first dosing up to 42 days post-dose
CHF10073 plasma Cmax (Maximum Plasma Concentration) | From first dosing up to 42 days post-dose

SECONDARY OUTCOMES:
CHF10073 plasma AUCinf (Area Under the Curve from time 0 Extrapolated to Infinity) | From first dosing up to 42 days post-dose
CHF10073 plasma tmax (Time to Maximum Plasma Concentration) | From first dosing up to 42 days post-dose
CHF10073 plasma elimination half-life | From first dosing up to 42 days post-dose
CHF10073 plasma apparent clearance (CL/F) | From first dosing up to 42 days post-dose
CHF10073 plasma apparent volume of distribution (Vz/F) | From first dosing up to 42 days post-dose
CHF10073 urine amount excreted (Ae) | Part 1, 2 and 4 : From first dosing up to 28 days post-dose
CHF10073 urine faction excreted (fe) | Part 1, 2 and 4: From first dosing up to 28 days post-dose
CHF10073 renal clearance (CLr) | Part 1, 2 and 4: From first dosing up to 28 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jelle Klein, MD, Principal Investigator — SGS Belgium
Locations (1):
- SGS Belgium NV Clinical Pharmacology Unit, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No